CLINICAL TRIAL: NCT02272777
Title: An Open-label Multi-center Study of Imatinib and Nilotinib in CAMN107ECN02 On-treatment Patients With Philadelphia Chromosome Positive Chronic Myelogenous Leukemia in Chronic Phase After the End of CAMN107ECN02 Core Study
Brief Title: A Study of Imatinib and Nilotinib in Patients With Chronic Myelogenous Leukemia in Chronic Phase
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107ECN02E1
Record Dates: First submitted 2014-10-21; First posted 2014-10-23 (Estimated); Results first posted 2019-08-19 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-07

CONDITIONS: Leukemia
Keywords: Nilotinib; AMN107; Tasigna; Imatinib; STI571; Gleevec/Glivec; BCR-ABL Positive; Philadelphia chromosome positive (Ph+) chronic myelogenous leukemia in chronic phase (CML-CP); Chronic myelogenous leukemia; Chronic myeloid leukemia; Chronic myelocytic leukemia; Acute Lymphoblastic Leukemia (ALL) Philadelphia chromosome positive; Acute Lymphoid Leukemia; suboptimal molecular response
MeSH Terms: conditions — Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Imatinib Mesylate; nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Imatinib (Active Comparator): Eligible patients from imatinib arm in core study CAMN107ECN02 were enrolled into imatinib arm in this study. Patients in imatinib 400 mg daily arm received imatinib daily dose of 300 mg, 400 mg or 600 mg all at once every day.
  Interventions: Drug: Imatinib
- Nilotinib (Experimental): Eligible patients from nilotinib arm in core study CAMN107ECN02 were enrolled into imatinib arm in this study. Patients in nilotinib arm received 300 mg BID by mouth each morning and evening approximately 12 hours apart, or 400 mg QD.
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Imatinib — Imatinib 400mg QD，300mg QD or 600mg QD
  Other Names: STI571, Gleevec/Glivec
  Arms: Imatinib
Drug: Nilotinib — Nilotinib 300mg BID or 400mg QD
  Other Names: AMN107, Tasigna
  Arms: Nilotinib

SUMMARY:
The extension study followed the core study CAMN107ECN02 (NCT01275196). which is an open-label, two armed study. All patients enrolled in this extension study were able to benefit from the treatment given in CAMN107ECN02 per investigator's evaluation. Therefore, in this extension study patient continued treatment of the drug (imatinib or nilotinib) which they were taking at the end of CAMN107ECN02. Treatment arms in CAMN107ECN02 were retained. As long as EC approval and agreement from investigators were obtained, the selected sites for CAMN107ECN02 were applied in this extension study.

DETAILED DESCRIPTION:
Up to 230 patients who benefited from the core study treatment (imatinib or nilotinib), at Investigator's discretion, were enrolled into this extension study. The patients continued receiving the open-label drugs that they were taken by the end of core study. Treatment arms in the core study were retained. No crossover between the arms was allowed.

The extension study started from the first patient last dose date in the core study and ends at the time of nilotinib was commercially available in China as a first line treatment. Eligibility evaluations were given for each patient before the enrollment. Follow-up visits at a frequency of 6 months were required to report AE, SAE and pregnancy only. No efficacy data were collected in the extension study since full efficacy had already been analyzed in the core study.

ELIGIBILITY:
Key Inclusion Criteria

1. Patient is currently on treatment in the core study CAMN107ECN02
2. Patient who continues to derive benefit more than risk from the study treatment he/she takes in CAMN107ECN02, in the opinion of the investigator at the end of the study
3. Written informed consent must be obtained prior to enrolling in the extension study

Key Exclusion Criteria:

1. Progression to CML-AP or BC
2. Patient whose treatment assigned in CAMN107ECN02 is not appropriate any longer, per investigator's assessment.
3. History of non-compliance to medical regimens, or patients who are considered potentially unreliable and/or not cooperative.
4. Women who are (a) pregnant and(b) women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and at least 14 days after last dose of study medication. Highly effective contraception methods include:

   * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
   * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
   * Male sterilization (at least 6 months prior to screening). For female subjects on the study the vasectomized male partner should be the sole partner for that subject.
   * Combination of any two of the following (a+b or a+c, or b+c):

     1. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.
     2. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
     3. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2014-07-17 (Actual); Primary Completion 2017-01-30 (Actual); Study Completion 2017-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- China (10):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Tianjin, Tianjin Municipality
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Fuzhou
  - Novartis Investigative Site, Jinan
  - Novartis Investigative Site, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 13 centers in China.
Pre-assignment Details: Patients continued treatment of the drug they were taking at the end of CAMN107ECN02 (NCT01275196). The starting dose had to be the same as the last dose that was given in the core study. After this, dose was based on the investigator's judgment.
Period: Overall Study
Arm/Group | Imatinib | Nilotinib
Started (All enrolled subjects were included in the Safety Set) | 112 | 113
Completed | 108 | 109
Not Completed | 4 | 4
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Lost to Follow-up | 2 | 0
Not completed — Other | 2 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Set was the only analysis set for this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Imatinib | Nilotinib | Total
Number analyzed (Participants) | 112 | 113 | 225
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.3 (12.8) | 45.5 (12.7) | 44.4 (12.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 38 | 83
  Male | 67 | 75 | 142
Race/Ethnicity, Customized [Number; unit: Participants]
  Chinese | 112 | 113 | 225

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Clinically significant changes in laboratory values and vital signs were reported as AEs or SAEs, as appropriate. Only descriptive analysis.
Time Frame: From first dose of study treatment to 30 days after last dose of study treatment, up to 31 months
Measure: Count of Participants; unit: Participants
Arm/Group | Imatinib | Nilotinib
Number analyzed (Participants) | 112 | 113
Participants
  Adverse Events (AEs) | 82 | 84
  Serious Adverse Events (SAEs) | 1 | 3
  Fatal SAEs | 0 | 0
  AEs leading to drug discontinuation | 0 | 1
  AEs leading to dose adjustment/interruption | 17 | 17

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for the maximum duration of participants' treatment exposure up to 29.3 months, plus 30 days follow up period.
Arm/Group | Imatinib | Nilotinib
All-Cause Mortality (participants affected / at risk) | 0/112 | 0/113
Serious Adverse Events (participants affected / at risk) | 1/112 | 3/113
Other Adverse Events (participants affected / at risk) | 74/112 | 68/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib (N=112) | Nilotinib (N=113)
Enteritis (Gastrointestinal disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib (N=112) | Nilotinib (N=113)
Anaemia (Blood and lymphatic system disorders) | 9 | 4
Leukopenia (Blood and lymphatic system disorders) | 10 | 2
Neutropenia (Blood and lymphatic system disorders) | 6 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 7
Nausea (Gastrointestinal disorders) | 7 | 1
Asthenia (General disorders) | 15 | 10
Chest discomfort (General disorders) | 6 | 4
Influenza (Infections and infestations) | 6 | 1
Upper respiratory tract infection (Infections and infestations) | 9 | 7
Alanine aminotransferase increased (Investigations) | 4 | 9
Blood bilirubin increased (Investigations) | 2 | 24
Blood cholesterol increased (Investigations) | 3 | 11
Blood creatine phosphokinase increased (Investigations) | 7 | 2
Blood creatinine increased (Investigations) | 9 | 0
Blood glucose increased (Investigations) | 9 | 8
Blood phosphorus decreased (Investigations) | 10 | 4
Blood triglycerides increased (Investigations) | 12 | 17
High density lipoprotein decreased (Investigations) | 7 | 3
Lipase increased (Investigations) | 6 | 7
Low density lipoprotein increased (Investigations) | 1 | 7
Weight increased (Investigations) | 7 | 5
White blood cell count decreased (Investigations) | 10 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 7
Hypophosphataemia (Metabolism and nutrition disorders) | 7 | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 6
Memory impairment (Nervous system disorders) | 10 | 10
Anxiety (Psychiatric disorders) | 6 | 3
Insomnia (Psychiatric disorders) | 2 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 5
Skin discolouration (Skin and subcutaneous tissue disorders) | 8 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-01-14): https://cdn.clinicaltrials.gov/large-docs/77/NCT02272777/SAP_000.pdf
  • Study Protocol (2014-05-27): https://cdn.clinicaltrials.gov/large-docs/77/NCT02272777/Prot_001.pdf